CLINICAL TRIAL: NCT01775176
Title: Effect of Weight and Insulin Sensitivity on Reproductive Function in Polycystic Ovary Syndrome: Studies in Skeletal Muscle and Adipose Tissue 'PULSE Ancillary Study'
Brief Title: Effect of Weight & Insulin Sensitivity on Reproductive Function in PCOS: Studies in Skeletal Muscle & Adipose
Acronym: PULSE-A
Status: Terminated | Type: Observational
Why Stopped: Parent Study stopped due to poor recruitment and enrollment
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Leanne Redman, Principle Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 11016-A
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS, Weight, Insulin Sensitivity, Reproductive Function
MeSH Terms: conditions — Polycystic Ovary Syndrome; Body Weight; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Skeletal Muscle Subcutaneous Adipose Tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Polycystic Ovary Syndrome: Overweight women with polycystic ovary syndrome. 20 - 40 years, inclusiveBody mass index ≥ 25kg/m2History of irregular menstrual cycles (fewer than 8 regular cycles in the past year)Clinical and/or biochemical androgen excess (Free androgen index>3.85 and/or hirsuitism rating ≥8)Anovulatory menstrual cycles (determined during screening)

SUMMARY:
The overall objective of this ancillary study is to obtain skeletal muscle and subcutaneous adipose tissue biopsies from women with polycystic ovary syndrome enrolled in the PULSE Study (NCT01482286).

DETAILED DESCRIPTION:
Muscle and adipose tissues will be appropriately collected and banked for future studies such as to measure expression of candidate genes involved with carbohydrate and fat oxidation and mitochondrial function by RT-PCR, protein content by western blot, enzyme activity by enzymatic assays and to perform functional studies under varying conditions (for example before and after treatment with insulin, testosterone, serum) to quantify insulin signaling and carbohydrate and fat oxidation in primary human cultures.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in PULSE NCT01482286

Exclusion Criteria:

* Withdraw from PULSE NCT01482286

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Overweight women with polycystic ovary syndrome.
  20 - 40 years, inclusive Body mass index ≥ 25kg/m2 History of irregular menstrual cycles (fewer than 8 regular cycles in the past year) Clinical and/or biochemical androgen excess (Free androgen index>3.85 and/or hirsuitism rating ≥8) Anovulatory menstrual cycles (determined during screening)
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Bio specimens for future research | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Leanne M Redman, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States